CLINICAL TRIAL: NCT06389214
Title: A Randomized, Double-Masked, Vehicle-Controlled Parallel Group Clinical Trial to Assess Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: A Clinical Trial to Assess the Efficacy and Safety of Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-030
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Disease
Keywords: dry eye; reproxalap
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) administered six times over two consecutive days (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution administered six times over two consecutive days (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered six times over two consecutive days
  Arms: Reproxalap Ophthalmic Solution (0.25%) administered six times over two consecutive days
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution administered six times over two consecutive days
  Arms: Vehicle Ophthalmic Solution administered six times over two consecutive days

SUMMARY:
A Randomized, Double-Masked, Vehicle-Controlled Parallel Group Clinical Trial to Assess Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

DETAILED DESCRIPTION:
Dry eye chamber challenge trial.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen to 70 years of age at the time of screening (either gender and any race)
* Ability to provide written informed consent
* Reported history of ocular discomfort associated with dry eye disease for at least 6 months prior to Visit 1
* Reported history of the use of eye drops for dry eye disease between 2 weeks to 6 months prior to Visit 1

Exclusion Criteria:

* Clinically significant slit lamp findings, intraocular pressure, and visual acuity findings at Visit 2 that may include active blepharitis, severe meibomian gland dysfunction, lid margin inflammation, glaucoma, ocular allergy, infection or any other disorder that, in the opinion of the Investigator, may interfere with trial conduct or assessments
* Diagnosis at Visit 1 of an ongoing ocular infection (bacterial, viral, or fungal), active ocular inflammation, or history of inflammatory disease that, in the opinion of the Investigator, could interfere with trial conduct or assessments
* Contact lens use within 7 days of Visit 1 or anticipated use of contact lenses during the trial
* Laser-assisted in situ keratomileusis (LASIK) surgery within 12 months of Visit 1 and/or planned ocular and/or lid surgeries during the trial or any other ocular surgery within 6 months of Visit 1
* Systemic corticosteroid or other immunomodulatory therapy (not including inhaled corticosteroids) within 60 days of Visit 1, or any planned immunomodulatory therapy during the trial
* Eye drop use within 2 weeks of Visit 1 and/or an unwillingness to discontinue any topical ophthalmic prescription or over-the-counter solutions, artificial tears, gels, or scrubs for the duration of the trial (excluding medications allowed for the conduct of the trial)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Ocular discomfort symptom score over 100 minutes in the dry eye chamber at Visit 2 and Visit 4 | From Day -14 to Day 2
  Measured using a 0 - 100 visual analog scale (VAS) where 0 is "no discomfort" and 100 is "maximal discomfort"

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Couroux, MD, Principal Investigator — Cliantha Research
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No